CLINICAL TRIAL: NCT01660438
Title: Prospective, Non-randomized, Observational Study of the Surgical Management of Suburethral Slings in Women With Stress Urinary Incontinence
Brief Title: Urethral Length Measurement in Women Undergoing Suburethral Sling Operative Procedure
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital, Frauenfeld (Other)
Responsible Party: Principal Investigator, Prof. Dr. Volker Viereck, Prof. Dr. Volker Viereck, Cantonal Hospital, Frauenfeld
Other Study IDs: TVT 112010
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence; Suburethral sling
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stress urinary incontinence: Stress urinary incontinence

SUMMARY:
This is a prospective, non-randomized, observational, multicenter study in which urethral length is measured in women with surgically-correctable stress urinary incontinence who undergo a suburethral sling operative procedure.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, observational, multicenter study in which urethral length is measured in women with surgically-correctable stress urinary incontinence who undergo a suburethral sling operative procedure. Data will be collected from preoperative urogynecological testing and medical histories. The urethral length will be measured intraoperatively using scaled catheters. Outcome data, including the development of postoperative complications, will be collected at several time intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has objective, demonstrable signs of stress urinary incontinence (SUI), including patients with intrinsic sphincter deficiency (ISD). Objective testing includes: standing stress test, urodynamics evaluation or pad test.
2. Patient is age 18 or older.
3. Patient agrees to participate in the study, including completion of all study-related procedures and evaluations, and documents this agreement by signing the Institutional Review Board/Ethics Committee-approved informed consent form.
4. Patient is able to fill in all questionnaires (based on judgment of investigator)

Exclusion Criteria:

1. Patient has an associated or suspected neurological disease.
2. Patient has an active lesion or present injury to perineum or urethra.
3. Patient has a urethral obstruction.
4. Patient has significant pelvic organ prolapse (Grade III/IV) requiring surgical treatment.
5. Patient has current urinary tract infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who have surgically-correctable stress urinary incontinence and undergo a suburethral sling operative procedure.
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2010-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Cure rate | 3 months
  Patients are classified as 'cured' if the postoperative cough test is negative, the 1-hour pad test is negative (less than 2 g) and the degree of subjective suffering improves to over 90% (VAS score of 0 or 1). All other patients are classified as therapeutic 'failures', even though they may experience marked improvement in one of the parameters compared with their preoperative status.

SECONDARY OUTCOMES:
Pelvic floor sonography | Pre-operation, day 1 and 3 months
Residual urine | Pre-operation, day 1 and 3 months
Pad test | Pre-operation and 3 months
Urethral length measurement | Intra-operation
  Urethral length will be measured using scaled catheters.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Viereck, Prof. Dr., Principal Investigator — Cantonal Hospital, Frauenfeld
Locations (3):
- Department of Gynecology and Obstetrics, Lutheran Hospital Hagen-Haspe, Hagen, Germany
- Szpital im M. Madurowicza, Lodz, Poland
- Blasenzentrum, Cantonal Hospital, Frauenfeld, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided